CLINICAL TRIAL: NCT07253805
Title: Plasma and Tissue Concentration of Cefazolin in Preoperative Prophylaxis in Patients Undergoing Bariatric Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Fondation IUCPQ (Other)
Responsible Party: Principal Investigator, François Julien, General and Bariatric Surgeon, and Clinical Researcher, MD., Laval University
Other Study IDs: CER 21626, 2019-3053
Record Dates: First submitted 2025-11-13; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Bariatric Sleeve Gastrectomy; Cefazolin
Keywords: Cefazolin; Ancef; Bariatric surgery; Sleeve; gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen tissue (dermis and adipose tissue) and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clindamycin group/control: A control group of 10 patients undergoing sleeve gastrectomy at the Quebec Heart and Lung Institute, who have not been exposed to cefazolin due to penicillin allergy, will be recruited to validate the analytical method. During surgery, biopsies of adipose and dermal tissue and blood samples will be collected. No other antibiotic or medications will be administered to these patients.
- Ancef group: Sixty patients will be recruited for the study, with 20 patients assigned to each weight category. Recruitment will take place during the preoperative consultation at the bariatric surgery clinic. All patients expressing interest will be included, provided they do not meet any exclusion criteria (convenience sampling). During surgery, biopsies of adipose and dermal tissue and blood samples, will be collected. No additional antibiotics or medications will be administered to these patients.

SUMMARY:
This study investigates whether current cefazolin dosing guidelines for obese patients-2 g IV for those <120 kg and 3 g IV for those ≥120 kg-achieve adequate plasma and tissue concentrations (≥8 mg/L) for effective surgical prophylaxis. While several retrospective and prospective studies suggest that a 2 g dose may be sufficient regardless of weight, findings are inconsistent and often rely solely on plasma concentrations. Given that tissue concentration at the site of action is a more relevant pharmacokinetic marker, the study emphasizes the need to measure cefazolin levels in adipose tissue. Previous research using microdialysis has shown reduced tissue distribution in obese patients, potentially warranting higher doses. The study also highlights variability in defining the minimum inhibitory concentration (MIC) required for prophylaxis, noting that 8 mg/L is often considered the threshold for Enterobacteriaceae. Ultimately, the study aims to clarify whether current dosing achieves effective antibiotic levels across different weight categories, with a focus on tissue concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI ≥ 35 kg/m²
* Undergo bariatric surgery (sleeve gastrectomy) via laparoscopy

Exclusion Criteria:

* Under 18 years of age
* Weight over 180 kg
* Penicillin allergy
* Pregnant or breastfeeding women
* Chronic kidney disease (eGFR < 60 ml/min according to the Cockcroft-Gault equation)
* Liver cirrhosis
* Intraoperative blood loss ≥ 1 liter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults undergoing bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) of Cefazolin in Plasma, Adipose Tissue, and Dermal Tissue | During surgery
  AUC of cefazolin will be measured in plasma, adipose tissue, and dermal tissue at 0 minutes, 30 minutes, and at the end of surgery following administration according to current dosing guidelines.
  Unit of Measure:
  mg·min/L

SECONDARY OUTCOMES:
Proportion of Patients Achieving Cefazolin Tissue Concentrations ≥ 8 mg/L | During surgery
  Proportion of patients with adipose and dermal tissue concentrations of cefazolin ≥ 8 mg/L at any time point (0 min, 30 min, end of surgery), based on the MIC for Enterobacteriaceae.
  Unit of Measure:
  Percentage of patients (%)
Proportion of Patients Achieving Cefazolin Plasma Concentrations ≥ 2 mg/L | During surgery
  Proportion of patients with plasma concentrations of cefazolin ≥ 2 mg/L at each time point (0 min, 30 min, end of surgery), based on the MIC for methicillin-sensitive Staphylococcus aureus (MSSA).
  Unit of Measure:
  Percentage of patients (%)
Comparison of Cefazolin Concentrations Across Weight Categories | During surgery
  Comparison of plasma and tissue concentrations of cefazolin across weight categories (<120 kg, 120-149 kg, ≥150 kg) to identify potential underexposure in higher weight groups.
  Unit of Measure:
  Mean concentration (mg/L)
Tissue-to-Plasma Concentration Ratio of Cefazolin | During surgery
  Ratio of cefazolin concentration in tissue to plasma at each time point to assess distribution efficiency.
  Unit of Measure:
  Ratio (unitless)
Time Above MIC (T>MIC) for Cefazolin in Plasma and Tissue | During surgery
  Duration (in minutes) that cefazolin concentrations remain above MIC in plasma and tissue compartments, if additional time points are available.
  Unit of Measure:
  Minutes

OTHER OUTCOMES:
Screening and Eligibility Verification Through Demographic and Clinical Data | Preoperative period
  Participants will be evaluated during preoperative consultation by a bariatric surgeon. If eligible, informed consent will be obtained. Demographic and clinical data will be collected to confirm inclusion criteria:
  * Height (cm)
  * Weight at recruitment (kg)
  * BMI at recruitment (kg/m²)
  * Allergy status to penicillin
  Blood samples will confirm:
  * Absence of liver cirrhosis
  * Absence of chronic kidney disease (eGFR < 60 mL/min based on Cockcroft-Gault equation)
Demographic Data Collected Before Surgery for Eligibility Assessment | preoperative period
  Prior to the start of surgery, demographic data will be collected to confirm participant eligibility according to inclusion criteria and establish baseline characteristics.
  Data collected:
  * Age (years)
  * Weight at admission (kg); will be used to determine the appropriate prophylactic dose of cefazolin.
  * Body Mass Index (BMI) at admission (kg/m²)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Not applicable for this study

REFERENCES:
- [Result] Larkin M. Will India's medical sites learn from the US experience? Lancet. 2001 Jan 13;357(9250):155. doi: 10.1016/S0140-6736(05)71200-9. No abstract available. PMID 11197437
- [Result] Nicoli S, Santi P. Assay of amikacin in the skin by high-performance liquid chromatography. J Pharm Biomed Anal. 2006 Jun 7;41(3):994-7. doi: 10.1016/j.jpba.2005.12.029. Epub 2006 Feb 8. PMID 16466885
- [Result] Signs SA, File TM, Tan JS. High-pressure liquid chromatographic method for analysis of cephalosporins. Antimicrob Agents Chemother. 1984 Nov;26(5):652-5. doi: 10.1128/AAC.26.5.652. PMID 6517553
- [Result] Waltrip T, Lewis R, Young V, Farmer M, Clayton S, Myers S, Gray LA Jr, Galandiuk S. A pilot study to determine the feasibility of continuous cefazolin infusion. Surg Infect (Larchmt). 2002 Spring;3(1):5-9. doi: 10.1089/109629602753681104. PMID 12593694
- [Result] Chen X, Brathwaite CE, Barkan A, Hall K, Chu G, Cherasard P, Wang S, Nicolau DP, Islam S, Cunha BA. Optimal Cefazolin Prophylactic Dosing for Bariatric Surgery: No Need for Higher Doses or Intraoperative Redosing. Obes Surg. 2017 Mar;27(3):626-629. doi: 10.1007/s11695-016-2331-9. PMID 27520693
- [Result] Liu P, Muller M, Derendorf H. Rational dosing of antibiotics: the use of plasma concentrations versus tissue concentrations. Int J Antimicrob Agents. 2002 Apr;19(4):285-90. doi: 10.1016/s0924-8579(02)00024-9. PMID 11978499
- [Result] Hites M, Deprez G, Wolff F, Ickx B, Verleije A, Closset J, Loi P, Prevost J, Taccone FS, Racape J, Cotton F, Jacobs F. Evaluation of total body weight and body mass index cut-offs for increased cefazolin dose for surgical prophylaxis. Int J Antimicrob Agents. 2016 Dec;48(6):633-640. doi: 10.1016/j.ijantimicag.2016.08.019. Epub 2016 Oct 5. PMID 28128093
- [Result] van Kralingen S, Taks M, Diepstraten J, van de Garde EM, van Dongen EP, Wiezer MJ, van Ramshorst B, Vlaminckx B, Deneer VH, Knibbe CA. Pharmacokinetics and protein binding of cefazolin in morbidly obese patients. Eur J Clin Pharmacol. 2011 Oct;67(10):985-92. doi: 10.1007/s00228-011-1048-x. Epub 2011 Apr 16. PMID 21499760
- [Result] Ho VP, Nicolau DP, Dakin GF, Pomp A, Rich BS, Towe CW, Barie PS. Cefazolin dosing for surgical prophylaxis in morbidly obese patients. Surg Infect (Larchmt). 2012 Feb;13(1):33-7. doi: 10.1089/sur.2010.097. Epub 2012 Feb 8. PMID 22316145
- [Result] Unger NR, Stein BJ. Effectiveness of pre-operative cefazolin in obese patients. Surg Infect (Larchmt). 2014 Aug;15(4):412-6. doi: 10.1089/sur.2012.167. Epub 2014 May 13. PMID 24824510
- [Result] Pories WJ, van Rij AM, Burlingham BT, Fulghum RS, Meelheim D. Prophylactic cefazolin in gastric bypass surgery. Surgery. 1981 Aug;90(2):426-32. PMID 7020141
- [Result] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists; Infectious Disease Society of America; Surgical Infection Society; Society for Healthcare Epidemiology of America. Clinical practice guidelines for antimicrobial prophylaxis in surgery. Am J Health Syst Pharm. 2013 Feb 1;70(3):195-283. doi: 10.2146/ajhp120568. No abstract available. PMID 23327981
- [Result] Shabanzadeh DM, Sorensen LT. Laparoscopic surgery compared with open surgery decreases surgical site infection in obese patients: a systematic review and meta-analysis. Ann Surg. 2012 Dec;256(6):934-45. doi: 10.1097/SLA.0b013e318269a46b. PMID 23108128
- [Result] Peppard WJ, Eberle DG, Kugler NW, Mabrey DM, Weigelt JA. Association between Pre-Operative Cefazolin Dose and Surgical Site Infection in Obese Patients. Surg Infect (Larchmt). 2017 May/Jun;18(4):485-490. doi: 10.1089/sur.2016.182. Epub 2016 Dec 1. PMID 27906601
- [Result] Chopra T, Zhao JJ, Alangaden G, Wood MH, Kaye KS. Preventing surgical site infections after bariatric surgery: value of perioperative antibiotic regimens. Expert Rev Pharmacoecon Outcomes Res. 2010 Jun;10(3):317-28. doi: 10.1586/erp.10.26. PMID 20545596
- [Result] Freeman JT, Anderson DJ, Hartwig MG, Sexton DJ. Surgical site infections following bariatric surgery in community hospitals: a weighty concern? Obes Surg. 2011 Jul;21(7):836-40. doi: 10.1007/s11695-010-0105-3. PMID 20198452
- [Result] Christou NV, Jarand J, Sylvestre JL, McLean AP. Analysis of the incidence and risk factors for wound infections in open bariatric surgery. Obes Surg. 2004 Jan;14(1):16-22. doi: 10.1381/096089204772787239. PMID 14980028
- [Result] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621
- [Result] Buchwald H, Oien DM. Metabolic/bariatric surgery worldwide 2011. Obes Surg. 2013 Apr;23(4):427-36. doi: 10.1007/s11695-012-0864-0. PMID 23338049
- [Result] Lim SS, Vos T, Flaxman AD, Danaei G, Shibuya K, Adair-Rohani H, Amann M, Anderson HR, Andrews KG, Aryee M, Atkinson C, Bacchus LJ, Bahalim AN, Balakrishnan K, Balmes J, Barker-Collo S, Baxter A, Bell ML, Blore JD, Blyth F, Bonner C, Borges G, Bourne R, Boussinesq M, Brauer M, Brooks P, Bruce NG, Brunekreef B, Bryan-Hancock C, Bucello C, Buchbinder R, Bull F, Burnett RT, Byers TE, Calabria B, Carapetis J, Carnahan E, Chafe Z, Charlson F, Chen H, Chen JS, Cheng AT, Child JC, Cohen A, Colson KE, Cowie BC, Darby S, Darling S, Davis A, Degenhardt L, Dentener F, Des Jarlais DC, Devries K, Dherani M, Ding EL, Dorsey ER, Driscoll T, Edmond K, Ali SE, Engell RE, Erwin PJ, Fahimi S, Falder G, Farzadfar F, Ferrari A, Finucane MM, Flaxman S, Fowkes FG, Freedman G, Freeman MK, Gakidou E, Ghosh S, Giovannucci E, Gmel G, Graham K, Grainger R, Grant B, Gunnell D, Gutierrez HR, Hall W, Hoek HW, Hogan A, Hosgood HD 3rd, Hoy D, Hu H, Hubbell BJ, Hutchings SJ, Ibeanusi SE, Jacklyn GL, Jasrasaria R, Jonas JB, Kan H, Kanis JA, Kassebaum N, Kawakami N, Khang YH, Khatibzadeh S, Khoo JP, Kok C, Laden F, Lalloo R, Lan Q, Lathlean T, Leasher JL, Leigh J, Li Y, Lin JK, Lipshultz SE, London S, Lozano R, Lu Y, Mak J, Malekzadeh R, Mallinger L, Marcenes W, March L, Marks R, Martin R, McGale P, McGrath J, Mehta S, Mensah GA, Merriman TR, Micha R, Michaud C, Mishra V, Mohd Hanafiah K, Mokdad AA, Morawska L, Mozaffarian D, Murphy T, Naghavi M, Neal B, Nelson PK, Nolla JM, Norman R, Olives C, Omer SB, Orchard J, Osborne R, Ostro B, Page A, Pandey KD, Parry CD, Passmore E, Patra J, Pearce N, Pelizzari PM, Petzold M, Phillips MR, Pope D, Pope CA 3rd, Powles J, Rao M, Razavi H, Rehfuess EA, Rehm JT, Ritz B, Rivara FP, Roberts T, Robinson C, Rodriguez-Portales JA, Romieu I, Room R, Rosenfeld LC, Roy A, Rushton L, Salomon JA, Sampson U, Sanchez-Riera L, Sanman E, Sapkota A, Seedat S, Shi P, Shield K, Shivakoti R, Singh GM, Sleet DA, Smith E, Smith KR, Stapelberg NJ, Steenland K, Stockl H, Stovner LJ, Straif K, Straney L, Thurston GD, Tran JH, Van Dingenen R, van Donkelaar A, Veerman JL, Vijayakumar L, Weintraub R, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams W, Wilson N, Woolf AD, Yip P, Zielinski JM, Lopez AD, Murray CJ, Ezzati M, AlMazroa MA, Memish ZA. A comparative risk assessment of burden of disease and injury attributable to 67 risk factors and risk factor clusters in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2224-60. doi: 10.1016/S0140-6736(12)61766-8. PMID 23245609
- [Result] Ng M, Fleming T, Robinson M, Thomson B, Graetz N, Margono C, Mullany EC, Biryukov S, Abbafati C, Abera SF, Abraham JP, Abu-Rmeileh NM, Achoki T, AlBuhairan FS, Alemu ZA, Alfonso R, Ali MK, Ali R, Guzman NA, Ammar W, Anwari P, Banerjee A, Barquera S, Basu S, Bennett DA, Bhutta Z, Blore J, Cabral N, Nonato IC, Chang JC, Chowdhury R, Courville KJ, Criqui MH, Cundiff DK, Dabhadkar KC, Dandona L, Davis A, Dayama A, Dharmaratne SD, Ding EL, Durrani AM, Esteghamati A, Farzadfar F, Fay DF, Feigin VL, Flaxman A, Forouzanfar MH, Goto A, Green MA, Gupta R, Hafezi-Nejad N, Hankey GJ, Harewood HC, Havmoeller R, Hay S, Hernandez L, Husseini A, Idrisov BT, Ikeda N, Islami F, Jahangir E, Jassal SK, Jee SH, Jeffreys M, Jonas JB, Kabagambe EK, Khalifa SE, Kengne AP, Khader YS, Khang YH, Kim D, Kimokoti RW, Kinge JM, Kokubo Y, Kosen S, Kwan G, Lai T, Leinsalu M, Li Y, Liang X, Liu S, Logroscino G, Lotufo PA, Lu Y, Ma J, Mainoo NK, Mensah GA, Merriman TR, Mokdad AH, Moschandreas J, Naghavi M, Naheed A, Nand D, Narayan KM, Nelson EL, Neuhouser ML, Nisar MI, Ohkubo T, Oti SO, Pedroza A, Prabhakaran D, Roy N, Sampson U, Seo H, Sepanlou SG, Shibuya K, Shiri R, Shiue I, Singh GM, Singh JA, Skirbekk V, Stapelberg NJ, Sturua L, Sykes BL, Tobias M, Tran BX, Trasande L, Toyoshima H, van de Vijver S, Vasankari TJ, Veerman JL, Velasquez-Melendez G, Vlassov VV, Vollset SE, Vos T, Wang C, Wang X, Weiderpass E, Werdecker A, Wright JL, Yang YC, Yatsuya H, Yoon J, Yoon SJ, Zhao Y, Zhou M, Zhu S, Lopez AD, Murray CJ, Gakidou E. Global, regional, and national prevalence of overweight and obesity in children and adults during 1980-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2014 Aug 30;384(9945):766-81. doi: 10.1016/S0140-6736(14)60460-8. Epub 2014 May 29. PMID 24880830
- See also: WHO- Obesity and overweight- May, 7, 2025 — https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT07253805/Prot_SAP_000.pdf